CLINICAL TRIAL: NCT04019912
Title: A Randomized Trial on the Novel Use of Treadmill Plus Music in Multiple Sclerosis Patients With Gate Impairnent
Brief Title: The Novel Use of Treadmill Plus Music in MS Patients Gate Rehabilitation
Acronym: SMUSIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, Medical Director, Neurologist, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRCCSME 5/19
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Interventional Study
Keywords: Gait rehabilitation; Rhythmic auditory stimulation; GaitTrainer3; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The study is a parallel-group randomized clinical trial using a double-blind study design. The enrolled patients will be randomly assigned to the 2 groups using an automated computerized randomization program. Patients will be informed about the research and will be asked to fill in the informed consent form. The patient's basic characteristics (age, sex, duration of the illness, marital status and educational background) will be recorded. Randomization will be performed using a randomization list, so patients will be randomized in a 1:1 ratio in the intervention or control group. The randomization list is blind to anyone involved in informing potential study participants.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study uses a single-blinded study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait Training plus music (Experimental): Patients will be randomly assigned to the rehabilitation group through gait trainer3 with Rhythmic Auditory Stimulation (RAS). All patients will undergo a complete clinical and neurophysiological evaluation at baseline. The training program consist of 45 minutes of treadmill training with RAS. The daily training program will be practiced once a day at the same time of day (from 9:00 am to 1:00 pm), five times a week for eight consecutive weeks. RAS treadmill sessions will be performed individually in the same position and under the supervision of physiotherapists with 2 years of RAS training.
  Interventions: Other: Gait Training plus music
- Traditional Gait Training (Active Comparator): Patients will be randomly assigned to the non-Rhythmic Auditory Stimulation (RAS) treadmill walking group. All patients will undergo a complete clinical and neurophysiological evaluation at baseline.The daily training program consist of 45 minutes of conventional gait training using a non-RAS treadmill. The daily training program will be practiced once a day at the same time of day (from 9:00 am to 1:00 pm), five times a week for eight consecutive weeks. Non-RAS treadmill sessions will be performed individually in the same position and under the supervision of physiotherapists.
  Interventions: Other: Traditional Gait Training

INTERVENTIONS:
Other: Gait Training plus music — GaitTrainer3 is a platform that integrates gait training via a treadmill and RAS. The device is indeed equipped with an instrumented deck that issues acoustic cues to determine the exact tempo and rhythm during gait training and visual real-time biofeedback to prompt patients to follow their gait pattern. In fact, the device provides online feedback, including step length, speed, and symmetry, to encourage patient progress and monitor patient performance. Patient footfalls were compared in real-time to the desired footfalls step by step and documented in a histogram.
  Other Names: GaitTrainer3
  Arms: Gait Training plus music
Other: Traditional Gait Training — The traditional training will be provided by a conventional treadmill.
  Arms: Traditional Gait Training

SUMMARY:
Multiple sclerosis (MS) is characterized by demyelination andaxonal loss of the central nervous system, which progressively results in neurologic dysfunction and is often accompanied by gaite limitations, reduced fitness, and increased risk of falls. Traditional exercises such as treadmill walking orstationary cycling can often be perceived as boring, because theseexercises usually involve repetitive, continuous movements. In recents years the positive effect of the auditory stimulus in the recovery of gait difficulties has been demonstrated in Parkinson's disease, however this methodology on MS patients has been poorly investigated. In addiction the neurophysiological mechanisms by which coupling steps with external auditory cues improves gait remain partially unclear. For this reason, our purpose is to investigate whether patients with MS, compared to the control group, may have improvements in motor and psychological well-being, through training with devices that integrate motor training with musical stimuli (Gait trainer).

DETAILED DESCRIPTION:
Although the number of studies and the extent of available evidence is greater in case of parkinsonism, there is also evidence of the effects of music-based interventions on supporting motor function and emotional well-being in people with multiple sclerosis. Interventions based on music can influence multiple functions. Recently it has been shown that coupling of auditory signals with motor training may be possible to form a rhythmic gait by dragging movement patterns, supporting the generation of better gait patterns; moreover, it can have effects on the rhythmic dragging; the commitment of automatic timing systems; movement planning, execution and learning; and an increase in motivation. Furthermore, this type of coupling has been shown to improve various gait parameters, including cadence, gait speed, stride length, gait time variability and pitch width.

The aim of our study is to evaluate the effectiveness of the treadmill training combined with RAS in terms of mobility, balance and gait parameters, patient's well-being.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of relapsing remitting MS according to Polman criteria;
* presence of gait impairment;
* absence of auditory deficits;
* EDSS <4.5;
* absence of clinical and/or neuroradiological MS relapse in the 3 months before enrolment;
* stable therapy in the last 3 months.

Exclusion criteria:

* presence of bone or joint disorders;
* history of severe cardiovascular, respiratory, auditory, and muscular-skeletal disease;
* other neurological conditions; and neurologic music therapy in the last 3 month;
* MS relapse in the 6 months before enrolment;
* Expanded Disability Status Scale (EDSS) > 4.5.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Ten-metre walking test | 3 months
  The 10 Metre Walk Test (10MWT) is a performance measure used to assess walking speed in metres per second over a short distance.
Timed up-and-go test | 3 months
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance

SECONDARY OUTCOMES:
Gait Quality Index | 3 months
  BTS GAITLAB supplies to the physician the quantitative information and objective data needed to identify and analyze walking and posture problems, load anomalies and muscle failure, which would not be measurable with normal clinical exams.
  The digital synchronization of different analysis tools helps to simultaneously compare, frame by frame, the patient's movements of limbs and muscles and force distribution on the surface during movement.
Multiple Sclerosis Quality of Life-54 | 3 months
  The Multiple Sclerosis Quality of Life-54 (MSQOL-54) is a multidimensional health-related quality of life measure, assessing the perception of physical and mental well-being. The instrument is composed of 54 items concerning 12 subscales, which form two scales relating to the physical and mental well-being. The score of the physical function scales, perceptions of health, energy/fatigue, role-physical limitations, pain, sexual function, social function, health distress, is added and corrected to obtain a score on the MSQUOL PHYSICAL HEALTH scale: a score above 50.0 indicates physical well-being. The score of the health distress scale, overall quality of life, emotional well-being, role limitations - emotional, cognitive function is summed and corrected to obtain a score on the scale MSQUOL MENTAL HEALTH: a score above 50.0 indicates mental well-being. The administration time is about 11-18 minutes, it can be completed by an interviewer or by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Rocco S Calabrò, MD, Study Director — IRCCS Centro Neurolesi
Locations (1):
- IRCCS Neurolesi, Messina, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Calabro RS, Naro A, Filoni S, Pullia M, Billeri L, Tomasello P, Portaro S, Di Lorenzo G, Tomaino C, Bramanti P. Walking to your right music: a randomized controlled trial on the novel use of treadmill plus music in Parkinson's disease. J Neuroeng Rehabil. 2019 Jun 7;16(1):68. doi: 10.1186/s12984-019-0533-9. PMID 31174570
- [Result] Shahraki M, Sohrabi M, Taheri Torbati HR, Nikkhah K, NaeimiKia M. Effect of rhythmic auditory stimulation on gait kinematic parameters of patients with multiple sclerosis. J Med Life. 2017 Jan-Mar;10(1):33-37. PMID 28255373
- [Result] Conklyn D, Stough D, Novak E, Paczak S, Chemali K, Bethoux F. A home-based walking program using rhythmic auditory stimulation improves gait performance in patients with multiple sclerosis: a pilot study. Neurorehabil Neural Repair. 2010 Nov-Dec;24(9):835-42. doi: 10.1177/1545968310372139. Epub 2010 Jul 19. PMID 20643882
- [Result] Ashoori A, Eagleman DM, Jankovic J. Effects of Auditory Rhythm and Music on Gait Disturbances in Parkinson's Disease. Front Neurol. 2015 Nov 11;6:234. doi: 10.3389/fneur.2015.00234. eCollection 2015. PMID 26617566